#### CONFIDENTIAL

# AMENDMENT #1 to STATISTICAL ANALYSIS PLAN FOR PROTOCOL 207213

A randomized, evaluator-blind, single-center and two-arm clinical study designed to evaluate the local tolerance and cosmetic efficacy of a topical skin care formulation in healthy female subjects with moderate to advanced photo-damaged facial skin who have undergone a 70% Glycolic Acid facial peel procedure

#### **BIOSTATISTICS DEPARTMENT**

#### GLAXOSMITHKLINE CONSUMER HEALTHCARE

PPD Principal Biostatistician, Biostatistics

inVentiv Health Clinical

Final Version 2.0

15<sup>th</sup> August 2017

| Timing for A | amendment: | ⊠ Before unblinding |
|---|---|---|
| | | After unblinding |
| SAP text: | | |
| Reason for A | amendment: | |
| 1) Descripti<br>Analysis | • | vidual scores at end of section 8.2 "Secondary |
| | ient data is not available for stats and frequency counts | r formal analyses for individual scores, swill be presented." |
| · - | on for a figure for dermator Analysis": | logist total score at end of section 8.1 |
| time with | "To visually inspect the treatment effect on dermatologist total score, a plot across<br>time with the raw means will be produced. The plot will display a different<br>symbol for each treatment group." | |
| | 3) Description for a figure for subject self-assessment total scores at end of section 8.2 "Secondary Analysis": | |
| "To visually inspect the treatment effect on subject self-assessment total scores, a plot across time with the raw means will be produced. The plot will display a different symbol for each treatment group." | | |
| The following | g listing will be produced f | for the topline summary: |
| Listing No. | Description | |
| 2.1 | Adverse Events – Safety | Population |

# **Appendix 2 List of Tables, Figures & Listings**

Reason for Amendment:

Additional figures will be created:

| Figures<br>No. | Table Title (including population) | Template |
|---|---|---|
| 9.3.2.1 | Subject Self-Assessment Scores – Total Score<br>- Safety Population | Figure 9.3.3.1 |
| 9.3.3.1 | Dermatologist Assessment Scores – Total<br>Score - Safety Population | Appendix 3 |

#### **Appendix 3 Templates for Tables, Figures & Listings**

#### Reason for Amendment:

Protocol No. 207213

Page x of y Program Run Date:xxxx

Figure 9.3.3.1

Dermatologist Assessment Scores - Total Score
Safety Population



- \* = Significant difference from baseline (p < 0.05)
- # = Significant difference from baseline between groups

Note: No statistical comparison between pre-procedure assessment and baseline total scores was made

Program file name xxxxxxxxxxxxxxxxx

Programmers Note: Figure to be created for Safety population. Same format for figures 9.3.2.1 Change the title, footnote and time points to match protocol.

# **Table of Contents**

| G | lossai | ry | 7 |
|----|--------------|--------------------------------------------|-------|
| 1 | Iı | ntroduction | 8 |
| 2 | O | Objectives | 8 |
| 3 | S | tudy Design | 8 |
| 4 | $\mathbf{S}$ | ample Size Determination | 9 |
| 5 | | ata Considerations | |
| | 5.1 | Analysis Populations | |
| | 5.2 | Subgroups/Stratification | |
| | 5.3 | Time Windows | |
| | 5.4 | Missing Data Handling | |
| 6 | D | emographics and Baseline Characteristics | |
| | 6.1 | Subject Disposition | 11 |
| | 6.2 | Demographics | 11 |
| 7 | T | reatment Compliance and Concomitant Medica | tions |
| | •• | ••••••••••••••••••••••••••••••••••••••• | 12 |
| | 7.1 | Treatment Compliance | 12 |
| | 7.2 | Concomitant Medications | 12 |
| 8 | A | nalysis | 12 |
| | 8.1 | Primary Analysis | 12 |
| | 8.2 | Secondary Analysis | 13 |
| | 8.3 | Other Analyses | 14 |
| 9 | $\mathbf{S}$ | afety Analysis | 14 |
| 10 | ) Iı | nterim Analysis | 15 |
| 11 | T | opline Summary | 15 |
| 12 | 2 C | Changes to Planned Analysis | 15 |
| 13 | R | deferences | 15 |
| A | ppen | dix 1 Study Schedule | 16 |

# Glossary

| AE | Adverse Event |
|--------|----------------------------------------------|
| CI | Confidence Interval |
| ITT | Intent-to-Treat |
| MedDRA | Medical Dictionary for Regulatory Activities |
| PP | Per Protocol |
| TEAE | Treatment Emergent Adverse Event |
| TEWL | Transepidermal Water Loss |

### 1 Introduction

This document describes the statistical methods and data presentations to be used in the summary and analysis of the final data from Protocol 207213.

# 2 Objectives

| Objective(s) | Endpoint(s) |
|---|---|
| Primary | |
| Assessment of the local tolerance of the test product in subjects who have undergone a 70% Glycolic Acid facial peel | Evaluator (Dermatologist) global assessment of tolerance |
| Secondary | |
| Assessment of skin recovery (change from baseline) over a period of 14 days in subjects | Combined (sum of) Evaluator (Dermatologist) scores for signs/symptoms of erythema, edema, desquamation and dryness |
| who have undergone a 70% Glycolic Acid facial peel | Individual Evaluator (Dermatologist) scores for erythema, edema, desquamation and dryness |
| | Combined (sum of) subject self-assessment scores for redness, pain, stinging/burning, itching, tightness and dryness |
| | Individual subject self-assessment scores for redness, pain, stinging/burning, itching, tightness and dryness |
| | Instrumental measurement of barrier function (Tewameter) and moisturisation (Corneometer) |
| | Subject global self-assessment |
| Assessment of skin recovery (change from baseline) between treatment groups. | All assessments and measurements listed above |

# 3 Study Design

• Evaluator-blind

- Single study center
- Parallel-group
- Healthy female subjects with moderate to advanced photo-damaged facial skin
- Single test product (Physiogel Calming Relief SPF 20 Cream) used in combination with commercial sunscreen ("washout product", Sunmax Sensitive SPF 50). All subjects were to use the commercial sunscreen and cleanser provided. Randomization was to two groups (test product, no test product) with product usage as shown in the table below:

| Randomized | Morning | Lunchtime* | Evening |
|------------|-----------------|--------------|-----------------|
| Group | | | |
| Group 1 | 1. Cleansing | 1. Sunscreen | 1. Cleansing |
| (Test | 2. Test Product | | 2. Test Product |
| product) | 3. Sunscreen | | |
| Group 2 | 1. Cleansing | 1. Sunscreen | 1. Cleansing |
| (No test | 2. Sunscreen | | |
| product) | | | |

<sup>\*</sup>Lunchtime application must be at least 3 hours after previous sunscreen application

## 4 Sample Size Determination

Approximately 130 healthy females within the ages of 30 and 60 years (inclusive) with Fitzpatrick Skin Classification II-IV and moderate to advanced photo-damaged skin will be screened to randomize 80 subjects to ensure approximately 60 subjects (30 subjects per group) successfully complete the study.

The sample size is based on clinical considerations and literature precedent [Narurkar, Schalka, Sulimovic, Kim]. With 30 subjects per treatment group, a change from baseline in Transepidermal Water Loss (TEWL) at least half the magnitude of the standard deviation (e.g. assume std=4 (ref. RH02030 after 2D strip), and 2.1 point mean change from baseline) can be detected at two-sided alpha=0.05 with 80% power.

#### 5 Data Considerations

#### 5.1 Analysis Populations

- All randomized subjects with at least one application of product in the test
  phase (i.e. test product for subjects randomized to receive test product (i.e. in
  Group 1) or sunscreen for subjects randomized not to receive test product (i.e.
  in Group 2)) will be included in the Safety population. Evaluator global
  assessment of tolerance, evaluator individual and subject individual
  assessments of tolerance and AE reporting will be based on the Safety
  population.
- All subjects in the safety population with at least one post-baseline efficacy (TEWL or corneometry) assessment will be included in the ITT population. All efficacy analyses will be based on the ITT population
- All subjects will be considered eligible for a Per Protocol (PP) population if
  they were randomized, received at least one application of product, had at
  least one post-procedure, post-treatment assessment available and no protocol
  violations deemed to affect <u>both</u> the primary tolerance endpoint (Evaluator
  global assessment) and the efficacy assessments (TEWL, corneometry).

Subjects with a protocol violation that is deemed to affect some, but not all, of the above 3 assessments will be part of the PP population, but their data will be excluded from the assessment at which the protocol violation occurred.

Violations that may lead to the exclusion of data for PP analysis include, but are not limited to, the following:

- Violation of inclusion or exclusion criteria at screening or baseline that may affect any of the above 3 assessments.
- o Non-compliance with assigned treatment regimen.
- Use of prohibited treatment or medication before or during the study, which
  it is felt will affect any of the above 3 assessments.

Violations will be documented in the Population Definitions document. The content of this document will be agreed upon between the Biostatistician and Clinical Research Scientist or designee post database lock but prior to breaking of the study blind.

A PP analysis will be performed for the Evaluator global assessment, TEWL and corneometry if there is more than 10% difference in the number of subjects

evaluable in either of the treatment groups for the ITT and PP populations.

#### 5.2 Subgroups/Stratification

There was no stratification in this study.

#### 5.3 Time Windows

All data will be accepted for analysis. Deviations from the scheduled nominal visit days are not expected. Any deviations will be noted in the deviation log and visits may be considered for exclusion from the Per Protocol population.

#### 5.4 Missing Data Handling

Missing data will not be imputed. All data available for dropouts will be considered in analyses.

### **6** Demographics and Baseline Characteristics

#### 6.1 Subject Disposition

The number of overall subjects screened and who screen failed will be presented with the number and percentage of subjects randomized and completing the study by product group.

The number and percentage of subjects, in the Safety, ITT and PP populations will be presented by product group and overall. The percentages will be based upon the total number of subjects randomized.

The number and percentage of subjects completing the study and not completing the study, including a breakdown of the reasons for not completing the study, will be presented by product group and overall. The percentages will be based upon the total number of subjects randomized

## 6.2 Demographics

Age will be summarized descriptively for each product group using means, medians and standard deviations. Race, gender, Fitzpatrick phototype and Glogau photoaging type will be summarized by product group using frequency counts and percentages.

# 7 Treatment Compliance and Concomitant Medications

### 7.1 Treatment Compliance

Treatment compliance (application of either the test product or sunscreen) will be assessed during the blinded data review meeting and a listing will be produced for evaluation of protocol violations only. No formal listing of these data will be produced for the study report.

#### 7.2 Concomitant Medications

Concomitant medications and concomitant non-drug treatment procedures will be assessed during the blinded data review meeting and a listing will be produced for evaluation of protocol violations only. No formal listing of these data will be produced for the study report.

### 8 Analysis

### 8.1 Primary Analysis

The primary evaluation of tolerance will be based on the Evaluator (Dermatologist) global assessment. The trial will be considered a success if the majority of subjects in the test product group have a favorable ("well tolerated") Evaluator global assessment score.

The Dermatologist will assess the local tolerance of the post-procedure skin care regimen in context of the expected effects of the procedure for each subject using the scale below and document the score on the eCRF. To make this assessment, the Dermatologist will draw on the total set of clinical and subject self-assessment data for each subject. The Dermatologist must be unaware of whether a subject was randomized to test product to protect the blind.

| Rating | Description |
|---|---|
| Well Tolerated | No clinically significant worsening of the expected signs/symptoms of the procedure. No new signs/symptoms manifest during product use. |
| Not Well Tolerated | Clear, clinically relevant worsening of the severity or frequency of expected signs/symptoms of the procedure and/or any occurrence of new, unexpected signs/symptoms during product use. |

Descriptive statistics (N, percentage, 95% confidence intervals) will be used to summarize the proportion of subjects in each product group with a favorable Evaluator global assessment of tolerance. The proportions will also be compared between product groups using Chi-square test, and difference in proportion and 95% confidence interval.

To visually inspect the treatment effect on dermatologist total score, a plot across time with the raw means will be produced. The plot will display a different symbol for each treatment group.

#### 8.2 Secondary Analysis

Efficacy measurements in this study will be based on changes from baseline in TEWL and Corneometer values at each timepoint. Both measurements will be assessed preprocedure and at Baseline (60±15 minutes post-procedure), 180 minutes post-procedure, 360 minutes post-procedure, and 1, 2, 3, 7 and 14 days post-procedure. The baseline for these measurements will be defined as the measurements made 60±15 minutes after the facial peel procedure, before any test product application.

Secondary assessments of local tolerance will be based on Evaluator (Dermatologist) and Subject self-assessment scores at each timepoint and reported adverse events. The baseline for these assessments will be defined as the assessments made 60±15 minutes after the facial peel procedure, before any test product application.

Evaluator and Subject assessment scores will be tabulated at each timepoint (Baseline (60±15 minutes post-procedure), 180 minutes post-procedure, and 1, 2, 3, 7 and 14 days post-procedure) for each product group descriptively as the number and percentage of subjects with each rating score for each assessment (none, mild, moderate or severe).

Changes from baseline in the Evaluator and Subject self-assessment and instrumental endpoints (TEWL and corneometry) will be tabulated by product group and timepoint and summarized descriptively using means, standard deviations and 95% confidence intervals and assessed for significance (different from zero) using t-tests or Wilcoxon signed rank tests dependent upon the distribution of the data.

Differences between product groups in the mean changes from baseline in Evaluator, and Subject self-assessment and instrumental endpoints will also be explored using t-tests or Wilcoxon rank sum tests at each timepoint and summarised using 95% confidence intervals.

If sufficient data is not available for formal analyses for individual scores, summary stats and frequency counts will be presented.

To visually inspect the treatment effect on subject self-assessment total scores, a plot

across time with the raw means will be produced. The plot will display a different symbol for each treatment group.

#### 8.3 Other Analyses

Subject global assessment of satisfaction evaluated at the last post-procedure follow-up visit (Day 22 – 14 days post-procedure) will be summarized by product group and tabulated for each rating descriptively using N and percentage of subjects. The ratings of "Very Satisfied" and "Satisfied" will also be combined and summarized descriptively (N, percent of subjects, 95% confidence intervals) by product group. The difference between product groups in the proportion of "Very Satisfied" and "Satisfied" subjects will also be presented with a 95% confidence interval for the difference and evaluated for a treatment difference via Chi-square test.

### 9 Safety Analysis

Adverse events will be tabulated by product group and listed for inspection.

As per Section 7.1 of the protocol, the following does not meet the definition of an adverse event:

- "Any clinically significant abnormal laboratory findings (if applicable) or
  other abnormal safety assessments which are associated with the underlying
  disease, unless judged by the investigator to be more severe than expected for
  the subject's condition."
- Therefore, the Dermatologist (erythema, edema, dryness, and desquamation) and Subject-self assessment (pain, stinging/burning, itching, tightness, redness, and dryness) grades will only be considered adverse events (AE) if they are scored as "Severe", **or** if the investigator judges them to be more severe than expected in context of the Glycolic Acid treatment procedure.

Treatment emergent AEs are defined as events that start on or after the first product application in the test phase.

AEs will be tabulated according to the current version of the MedDRA. Frequencies and percentages will be presented by product group and overall, for each system organ class, and for each preferred term. Summaries of treatment-emergent AEs (TEAEs), treatment-related TEAEs, TEAEs by severity and treatment-related TEAEs by severity.

Adverse events will be listed for the safety population and separately for the non-randomised subjects. Any serious AEs will also be listed.

### 10 Interim Analysis

Not Applicable

## 11 Topline Summary

The following tables will be produced for the topline summary:

| Table No. | Description |
|-----------|------------------------------------------------------------------|
| 9.1 | Subject Disposition by Treatment Group – All Screened Subjects |
| 9.3.1 | Summary of Evaluator Global Assessment Score – Safety Population |
| 9.3.4 | Summary of TEWL – Changes from Baseline – ITT Population |
| 9.3.5 | Summary of Corneometry – Changes from Baseline – ITT Population |
| 9.4.1 | Treatment-Emergent Adverse Events – Safety Population |
| Listing | Description |
| No. | |
| 2.1 | Adverse Events – Safety Population |

## 12 Changes to Planned Analysis

There are no changes to the protocol-planned statistical analyses however the analysis populations definitions were updated from the protocol (See Section 5.1 above). This is to update inclusion of one post baseline efficacy assessment for ITT population definition and clarification of what assessments will be analysed as per each population.

#### 13 References

None

# **Appendix 1 Study Schedule**

| | Visit 1<br>Day 1 | Visit 2<br>Day 2 | Visit 3 <sup>1</sup><br>Day 8 | Visit 4 <sup>1</sup><br>Day 9 | Visit 5 <sup>1</sup><br>Day 10 | Visit 6 <sup>1</sup><br>Day 11 | Visit 7 <sup>1</sup><br>Day 15 | Visit 8 <sup>1</sup><br>Day 22 |
|---|---|---|---|---|---|---|---|---|
| Procedure/ Assessment | Screening/<br>Washout | 1 Day After<br>Visit 1 | 6 Days after<br>Visit 2, Day<br>of Procedure | 1 Day after<br>Visit 3 | 1 Day after<br>Visit 4 | 1 Day after<br>Visit 5 | 4 Days after<br>Visit 6 | 7 Days after<br>Visit 7 |
| Informed Consent | X | | | | | | | |
| Demographics | X | | | | | | | |
| Medical History | X | | | | | | | |
| Current / Concomitant Medication | X | X | X | X | X | X | X | X |
| Adverse Events | | X | X | X | X | X | X | X |
| Continued Subject Eligibility | | X | X | X | X | X | X | X |
| Compliance (Diary review) <sup>2</sup> | | X | X | X | X | X | X | X |
| Fitzpatrick Skin Type Assessment (Appendix 2) | X | | | | | | | |
| Glogau Photoaging Type Assessment (Appendix 3) | X | | | | | | | |
| In/ExclusionCriteria | $\mathbf{X}^3$ | $X^4$ | $\mathbf{Y}^4$ | | | | | |
| Subject Eligibility | X | | • | | | | | |
| Study Material Sensitivity Test | <b>Y</b> <sup>5</sup> | | | | | | | |
| Subject Self-Assessment Sensitivity | V <sup>6</sup> | $\mathbf{v}^7$ | X | | | | | |
| Dermatologist Assessment Sensitivity | $X^6$ | $\mathbf{X}^7$ | X | | | | | |
| Exclusion Criteria 9 | X | | | | | | | |
| Subject Eligibility | X | X | X | | | | | |
| Subject Randomisation | | | X | | | | | |
| Instrumental Measurements Pre-Procedure | | | X | | | | | |
| Image capture (VISIA) Pre-Procedure | | | X | | | | | |
| Subject Self-Assessment Pre-Procedure | | | X | | | | | |
| Dermatologist Assessment Pre-Procedure | | | X | | | | | |
| Dermatological Procedure (Facial Peel) | | | $\mathbf{V}^8$ | | | | | |
| Dermatologist Assessment Post-Procedure,<br>Pre-Treatment (BASELINE) | | | X <sup>9</sup> | | | | | |
| Instrumental Measurements Post-<br>Procedure, Pre-Treatment (BASELINE) | | | X <sup>9</sup> | | | | | |
| Image capture (VISIA) Post-Procedure,<br>Pre-Treatment (BASELINE) | | | X <sup>9</sup> | | | | | |
| Subject Self-Assessment Post-Procedure,<br>Pre-Treatment (BASELINE) | | | X <sup>9</sup> | | | | | |
| Washout Products Weighing | X | X | X | X | X | X | X | X |
| Washout Products and Washout Diary<br>Dispensing | X | | | | | | | |

| Test Product Weighing | X | X | X | X | X | X |
|---|---|---|---|---|---|---|
| Test Product and Test Diary Dispensing,<br>Washout Diary return. | $X^{10}$ | | | | | |
| Supervised Test-Product Application Post-<br>Procedure | X <sup>11</sup> | | | | | |
| Instrumental Measurements Post-<br>Procedure, Post-Treatment <sup>12</sup> | X | X | X | X | X | X |
| Image capture (VISIA) Post-Procedure,<br>Post-Treatment | | X <sup>14</sup> | | | | X |
| Subject Self-Assessment Post-Procedure,<br>Post-Treatment <sup>13</sup> | X | X | X | X | X | X |
| Subject Global Self-Assessment | | | | | | X |
| Dermatologist Assessment Post-Procedure,<br>Post-Treatment <sup>13</sup> | X | X | X | X | X | X |
| Dermatologist Global Assessment of<br>Tolerance | | | | | | X |
| Supervised Test-Product Application <sup>15</sup> | | X | X | X | X | |
| Supervised Sunscreen Application <sup>16</sup> | | X | X | X | X | |
| Products and Test Diary Return | | | | | | X |
| Discharge from Study | | | | | | X |

- 1. For Visits 3-8, subjects will be instructed to cleanse their face at home using the cleanser provided and must not use any other product on their face, including the test product (Group I only) and sunscreen. Subjects will be instructed to bring the dispensed cleanser, sunscreen and test product (Group I only) with them to all visits. Subjects will be invited to the site in the morning (prior to 9 am) to avoid exposure to strong sunlight.
- 2. The Investigator or designee will review the diary to monitor and encourage compliance. Additional or missed product applications will be recorded as deviations. The Evaluator must be blind to diary review.
- 3. Exclusion Criteria 9 will not be included for this assessment. Exclusion criteria 9 is evaluated based on the results from the sensitivity test.
- 4. To include a review of the inclusion/exclusion criteria specified in Appendix 4. Subjects must be considered compliant with these inclusion/exclusion criteria in order to remain eligible for the study.
- 5. Peel regimen (70% Glycolic Acid facial peel solution, Bicarbonate Neutralizing Solution and Sunmax Sensitive SPF 50) to be applied to the volar forearm of each subject by a qualified dermatologist.
- 6. Assessments to be taken 45±15 minutes after completion of the study material sensitivity test product application is complete.
- 7. Assessments to be taken 24±4 hours after completion of the study material sensitivity test product application is complete.
- 8. 70% Glycolic Acid facial peel to be administered by a qualified dermatologist who must be blind to randomization. The Glycolic Acid treatment and neutralizing solution will be sourced commercially by the study site.
- 9. Assessments to be taken 60±15 minutes after completion of the facial peel procedure.
- 10. Only subjects randomised to Group I will be dispensed test product. Subjects in Group I and II will be dispensed different test diaries to reflect the difference in treatment allocation. The washout diary will be returned at the same time as test diary dispensing.
- 11. Test product application will occur immediately after the post-procedure, pre-treatment (Baseline) assessments are complete and under the supervision of the Investigator or designee to subjects in Group I, only. Subjects in Group II will not apply anything to their face. The Evaluator must be blind to test product application.
- 12. Measurements to be taken 180±15 minutes, 360±15 minutes, 24±4 hours, 48±4 hours, 72±4 hours, 168±4 hours and 336±4 hours after completion of the facial peel procedure. At Visit 3, there must be at least 30 minutes between test product application (Group I, only) and instrumental measurements.
- 13. Assessments to be taken 180±15 minutes, 24±4 hours, 48±4 hours, 72±4 hours, 168±4 hours and 336±4 hours after completion of the facial peel procedure.
- 14. Images to be captured 24±4 hours after completion of the facial peel procedure.

| | Test product application will be conducted under the supervision of the Investigator or designee to subjects in Group I, only. Subjects in Group II will not apply the test product to their face. |
|---|---|
| 16. | Sunscreen application will be conducted under the supervision of the Investigator or designee to all subjects. |

# **Appendix 2 List of Tables, Figures & Listings**

In all outputs, the treatment labels and order for presentation in tables and listings is:

- 1) Physiogel Calming Relief SPF 20 Cream
- 2) No Test Product

| Table No. | Table Title (including population) | Template |
|---|---|---|
| 9.1 | Subject Disposition by Treatment Group – All Screened Subjects | Appendix 3 |
| 9.2.1.1 | Demographics – ITT Population | Appendix 3 |
| 9.2.1.2 | Demographics – Safety Population | Table 9.2.1.1 |
| 9.2.1.3 | Demographics – PP Population (if needed) | Table 9.2.1.1 |
| 9.3.1 | Summary of Evaluator Global Assessment<br>Score – Safety Population | Appendix 3 |
| 9.3.2.1 | Summary of Subject Self-Assessment Scores – Individual Assessments - Safety Population | Table 9.3.3.1 |
| 9.3.2.2.1 | Summary of Subject Self-Assessment Scores –<br>Total Score - Changes from Baseline – Safety<br>Population | Table 9.3.3.2.1 |
| 9.3.2.2.2 | Summary of Subject Self-Assessment Scores –<br>Pain Score - Changes from Baseline - Safety<br>Population | Table 9.3.3.2.1 |
| 9.3.2.2.3 | Summary of Subject Self-Assessment Scores – Stinging/Burning Score - Changes from Baseline - Safety Population | Table 9.3.3.2.1 |
| 9.3.2.2.4 | Summary of Subject Self-Assessment Scores – Itching Score - Changes from Baseline - Safety Population | Table 9.3.3.2.1 |
| 9.3.2.2.5 | Summary of Subject Self-Assessment Scores –<br>Tightness Score - Changes from Baseline -<br>Safety Population | Table 9.3.3.2.1 |

| 9.3.2.2.6 | Summary of Subject Self-Assessment Scores – Redness Score - Changes from Baseline - Safety Population | Table 9.3.3.2.1 |
|---|---|---|
| 9.3.2.2.7 | Summary of Subject Self-Assessment Scores – Dryness Score - Changes from Baseline - Safety Population | Table 9.3.3.2.1 |
| 9.3.3.1 | Summary of Dermatologist Assessment Scores - Individual Assessments – Safety Population | Appendix 3 |
| 9.3.3.2.1 | Summary of Dermatologist Assessment Scores – Total Score - Change from Baseline – Safety Population | Appendix 3 |
| 9.3.3.2.2 | Summary of Dermatologist Assessment Scores – Erythema Score - Changes from Baseline - Safety Population | Table 9.3.3.2.1 |
| 9.3.3.2.3 | Summary of Dermatologist Assessment Scores - Dryness Score - Changes from Baseline - Safety Population | Table 9.3.3.2.1 |
| 9.3.3.2.4 | Summary of Dermatologist Assessment Scores - Desquamation Score - Changes from Baseline - Safety Population | Table 9.3.3.2.1 |
| 9.3.3.2.5 | Summary of Dermatologist Assessment Scores – Edema Score - Changes from Baseline - Safety Population | Table 9.3.3.2.1 |
| 9.3.4 | Summary of TEWL – Changes from Baseline – ITT Population | Table 9.3.3.2.1 |
| 9.3.4.1 | Summary of TEWL – Changes from Baseline – PP Population (if needed) | Table 9.3.3.2.1 |
| 9.3.5 | Summary of Corneometry – Changes from Baseline – ITT Population | Table 9.3.3.2.1 |
| 9.3.5.1 | Summary of Corneometry – Changes from Baseline – PP Population (if needed) | Table 9.3.3.2.1 |
| 9.3.6 | Summary of Subject Global Satisfaction – ITT Population | Appendix 3 |
| 9.4.1 | Treatment-Emergent Adverse Events – Safety Population | Appendix 3 |

| 9.4.2 | Treatment-Emergent Treatment-Related | 9.4.1 |
|-------|--------------------------------------|------------|
| | Adverse events – Safety Population | |
| 9.4.3 | Treatment-Emergent Adverse Events by | Appendix 3 |
| | Severity – Safety Population | |
| 9.4.4 | Treatment-Emergent Treatment-Related | 9.4.3 |
| | Adverse Events by Severity – Safety | |
| | Population | |

| Figures<br>No. | Table Title (including population) | Template |
|---|---|---|
| 9.3.2.1 | Subject Self-Assessment Scores – Total Score<br>- Safety Population | Figure 9.3.3.1 |
| 9.3.3.1 | Dermatologist Assessment Scores – Total<br>Score - Safety Population | Appendix 3 |

| Listing | Listing Title (including population) | Template |
|---------|------------------------------------------|------------|
| No. | | |
| 2.1 | Adverse Events – Safety Population | Appendix 3 |
| 2.2 | Adverse Events – Non-randomised Subjects | 2.1 |
| 2.3 | Serious Adverse Events | 2.1 |
| 2.4 | Randomisation Details | Appendix 3 |

**Appendix 3 Templates for Tables, Figures & Listings** 

Table 9.1
Subject Disposition by Treatment Group
All Screened Subjects

All Screened Subjects (N=xxx)

| | Physic | gel Calming Reli | ef | | | |
|---|---|---|---|---|---|---|
| | SP | F 20 Cream | No | Test Product | Overal | 1 |
| | N (% | ) | N ( | %) | N (%) | |
| TOTAL SUBJECTS SCREENED | | | | | XXX | |
| SUBJECTS NOT RANDOMIZED | | | | | xxx | |
| DID NOT MEET STUDY CRITERIA | | | | | XXX | (xx.x) |
| ADVERSE EVENT | | | | | Xxx | (xx.x) |
| LOST TO FOLLOW UP | | | | | XXX | (xx.x) |
| PROTOCOL VIOLATION | | | | | Xxx | (xx.x) |
| WITHDRAWAL OF CONSENT | | | | | Xxx | (xx.x) |
| OTHER | | | | | Xxx | (xx.x) |
| SUBJECTS RANDOMIZED | xxx | | xxx | | xxx | |
| COMPLETED STUDY | XXX | (xx.x) | XXX | (xx.x) | XXX | (xx.x) |
| DID NOT COMPLETE STUDY | XXX | (xx.x) | xxx | (xx.x) | XXX | (xx.x) |
| DID NOT MEET STUDY CRITERIA | XXX | (xx.x) | XXX | (xx.x) | XXX | (xx.x) |
| ADVERSE EVENT | XXX | (xx.x) | XXX | (xx.x) | XXX | (xx.x) |
| LOST TO FOLLOW-UP | XXX | (xx.x) | XXX | (xx.x) | XXX | (xx.x) |
| PROTOCOL VIOLATION | XXX | (xx.x) | XXX | (xx.x) | XXX | (xx.x) |
| WITHDRAWAL OF CONSENT | XXX | (xx.x) | XXX | (xx.x) | XXX | (xx.x) |
| OTHER | XXX | (xx.x) | XXX | (xx.x) | xxx | (xx.x) |
| TT POPULATION | xxx | (xx.x) | xxx | (xx.x) | xxx | (xx.x) |
| SAFETY POPULATION | XXX | (xx.x) | xxx | (xx.x) | XXX | (xx.x) |
| PP POPULATION | xxx | (xx.x) | xxx | (xx.x) | XXX | (xx.x) |

Program file name xxxxxxxxxxxxxxxxxxxxx

Programming note: For categories under 'Subjects Not Randomised' percentages will be calculated using the number of 'All Screened Subjects' as the denominator. Percentages under the 'Subjects Randomised' categories will be computed using number of subjects randomised as the denominator.

Table 9.2.1.1 Demographics ITT Population

ITT Population (N=xxx)

| SEX N (%) FEMALE RACE N (%) AMERICAN INDIAN OR ALASKA NATIVE | SPF 2<br>(N=:<br>xx | O Cream (xx.x) | No Te<br>(N=x | st Product<br>x) | Overa<br>(N=x | |
|---|---|---|---|---|---|---|
| FEMALE RACE N (%) AMERICAN INDIAN OR ALASKA NATIVE | xx | | | x) | (N=x | xx) |
| FEMALE RACE N (%) AMERICAN INDIAN OR ALASKA NATIVE | | (xx.x) | XX | | | |
| RACE N (%) AMERICAN INDIAN OR ALASKA NATIVE | | (xx.x) | XX | | | |
| AMERICAN INDIAN OR ALASKA NATIVE | xx | | | (xx.x) | XX | (xx.x) |
| | XX | | | | | |
| | | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| ASIAN | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| BLACK OR AFRICAN AMERICAN | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| WHITE | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| MULTIPLE | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| AGE (YEARS) | | | | | | |
| N | XX | | XX | | XX | |
| MEAN | XX. | X | XX. | X | XX. | X |
| SD | XX. | XX | XX. | XX | XX. | XX |
| MEDIAN | XX. | x | XX. | X | XX. | X |
| MINIMUM | XX | | XX | | XX | |
| MAXIMUM | XX | | XX | | xx | |
| FITPATRICK PHOTOTYPE N (%) | | | | | | |
| I | XX | (xx.x) | | | | • |
| II | XX | (xx.x) | | | | |
| III | XX | (xx.x) | | | | |
| IV | | | | | | |
| V | | | | | | |
| VI | | | | | | |
| GLOGAU PHOTOTYPE N (%) | | | | | | |
| Ī | XX | (xx.x) | | | | • |
| II | XX | (xx.x) | | | | |
| III | XX | (xx.x) | | | | |
| IV | | | | | | |
| Program file name xxxxxxxxxxxxxxxxxx | | | | | | |

# Table 9.3.1 Summary of Evaluator Global Assessment Score Safety Population

Safety Population (N=xx)

| | Physiogel Calming Relief | No Test Product |
|---|---|---|
| | SPF20 Cream | |
| N | xx | XX |
| Missing | XX (XX%) | XX (XX%) |
| Product Regimen was Well Tolerated | XX (XX%) | XX (XX%) |
| Product Regimen was Not Well Tolerated | XX (XX%) | XX (XX%) |
| 95% Confidence Interval for Proportion Well | (XX.X%, XX.X%) | (XX.X%, XX.X%) |
| Tolerated | | |
| Difference in Proportions Well Tolerated (95% | XX% (XX.X - | XX.X) |
| Confidence Interval) | | |
| Chi-Square P-Value | x.xxx | |

Percentages based on the total number of subjects per product group.

Program file name xxxxxxxxxxxxxxxxxx

Table 9.3.3.2.1

Summary of Dermatologist Assessments - Total Score®- Changes from Baseline
Safety Population

Safety Population (N=xx)

| Timepoint | | Physiogel Calming Relief | No Test Product |
|---|---|---|---|
| | | SPF 20 Cream | |
| Pre-Procedure Assessment | N | XX | XX |
| | Missing | XX | XX |
| | Mean | X.XX | X.XX |
| | SD | x.xxx | X.XXX |
| | 95%CI | x.xx, x.xx | X.XX, X.XX |
| Baseline* | N | XX | XX |
| | Missing | XX | XX |
| | Mean | X.XX | X.XX |
| | SD | x.xxx | X.XXX |
| | 95%CI | x.xx, x.xx | X.XX, X.XX |
| 180 Minutes Post-Procedure | N | XX | XX |
| | Missing | XX | XX |
| | Mean | X.XX | X.XX |
| | SD | x.xxx | X.XXX |
| | 95%CI | x.xx, x.xx | X.XX, X.XX |
| Change from Baseline at 180 | N | xx | XX |
| Minutes | Missing | xx | XX |
| | Mean | X.XX | X.XX |
| | SD | x.xxx | X.XXX |
| | 95%CI | x.xx, x.xx | X.XX, X.XX |

| | P-Value <sup>#</sup> | X.XXX | X.XXX |
|---|---|---|---|
| Difference between Groups at | Difference | X.XX (X.XX, X.XX) | |
| 180 Minutes | (95%CI) | | |
| | P-Value <sup>\$</sup> | X.XXX | |

Program file name xxxxxxxxxxxxxxxxxxx

Programmers Note: Continue table for each timepoint. Same format for Tables 9.3.2.2.x, 9.3.3.2.x, 9.3.4 and 9.3.5 - Change the title, footnote and timepoints to match protocol.

Total score=sum of Erythema, Dryness, Desquamation/Peeling and Edema individual scores.

 P-value from t-test or Wilcoxon signed rank test compared to zero.

 P-value from t-test or Wilcoxon rank sum test.

 Baseline score is assessed 60 minutes post-procedure and prior to any test product application.

# Table 9.3.3.1 Summary of Dermatologist Assessments - Individual Assessments Safety Population

Safety Population (N=xx)

| Physiogel Calming Relief SPF 20 Cream | No Test Product |
|---------------------------------------|-----------------|
| (N=xx) | (N=xx) |

| | Missing | None | Mild | Moderate | Severe | Total | Missing | None | Mild | Moderate | Severe | Total |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Erythema | | | | | | | | | | | | |
| Pre-procedure | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X |
| Baseline* Score | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X |
| 180 Min | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X |
| 1 Day | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X |
| 2 Days | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X |
| 3 Days | X(xx%) | X (xx%) | X (xx%) | X(xx%) | X(xx%) | X | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X |
| 7 Days | X(xx%) | X (xx%) | X (xx%) | X(xx%) | X(xx%) | X | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X |
| 14 Days | X(xx%) | X (xx%) | X (xx%) | X(xx%) | X(xx%) | X | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X |
| Dryness | | | | | | | | | | | | |
| Pre-procedure | ••• | | | | | | ••• | | | ••• | | |

Baseline\* Score

180 Min

1 Day

2 Days

3 Days

7 Days 14 Days

#### Desquamation

| Pre-procedure | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Baseline* Score | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X |
| 180 Min | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X |
| 1 Day | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X |
| 2 Days | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X |
| 3 Days | X (xx%) | X (xx%) | X (xx%) | X(xx%) | X(xx%) | X | X (xx%) | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X |
| 7 Days | X (xx%) | X (xx%) | X (xx%) | X(xx%) | X(xx%) | X | X (xx%) | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X |
| 14 Days | X (xx%) | X (xx%) | X (xx%) | X(xx%) | X(xx%) | X | X (xx%) | X(xx%) | X(xx%) | X(xx%) | X(xx%) | X |

#### Edema

Pre-procedure

Baseline\* Score

180 Min

1 Day

2 Days

3 Days

7 Days

14 Days

Percentages based on total number of subjects per product group.

Program file name xxxxxxxxxxxxxxxxxx

Programmer's note: Same format for table 9.3.2.1 (change assessments to match protocol).

 $<sup>^{\</sup>star}$  Baseline score is assessed 60 minutes post-procedure and prior to any test product application.

# Table 9.3.6 Summary of Subjects Global Assessment of Satisfaction Intent-to-Treat Population

ITT Population(N=xx)

| | Physiogel Calming Relief | No Test Product |
|---|---|---|
| | SPF 20 Cream (N=xx) | (N=xx) |
| N | XX | XX |
| Missing | XX (XX%) | XX (XX%) |
| Very Satisfied | XX (XX%) | XX (XX%) |
| Satisfied | XX (XX%) | XX (XX%) |
| - Total Satisfied and Very Satisfied | XX (XX%) | XX (XX%) |
| 95% Confidence Interval | XX.X%, XX.X% | XX.X%, XX.X% |
| Difference in Proportions Very Satisfied and | XX% (XX.X | - XX.X) |
| Satisfied (95% Confidence Interval) | | |
| Chi-Square P-Value | X.XX | X |
| Poorly Satisfied | XX (XX%) | XX (XX%) |
| Not at all Satisfied | XX (XX%) | XX (XX%) |

Percentages based on total number of subjects per product group.

Program file name xxxxxxxxxxxxxxxxxx

# Table 9.4.1 Treatment Emergent Adverse Events Safety Population

Safety Population (N=xx)

| | Physiogel Calming Relief<br>SPF 20 Cream<br>(N=XX) | No Test Product<br>(N=XX) | Overall<br>(N=XXX) |
|---|---|---|---|
| | n (%) nAE | n (%) nAE | n (%) nAE |
| NUMBER OF SUBJECTS WITH AT LEAST ONE AE | xx ( xx.x) xx | xx ( xx.x) xx | xx ( xx.x) xx |
| NUMBER OF SUBJECTS WITH NO AE | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| 50C1 | xx ( xx.x) xx | xx ( xx.x) xx | xx ( xx.x) xx |
| PT1 | xx ( xx.x) xx | xx (xx.x) xx | xx ( xx.x) xx |
| 50C2 | xx ( xx.x) xx | xx ( xx.x) xx | xx ( xx.x) xx |
| PT1 | xx ( xx.x) xx | xx ( xx.x) xx | xx ( xx.x) xx |

N (%) = Number (percent) of subjects

nAE = Number of adverse events

Program file name xxxxxxxxxxxxxxxxxx

Programmer's note: Same format for table 9.4.2

Table 9.4.3
Summary of Treatment Emergent Adverse Event by Severity
Safety Population

Safety Population (N=xx)

| System Organ Class | | Phys | siogel Cal | lming F | Relief | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Preferred Term | SPF 20 Cream | | | | | | No Test Product | | | | | |
| | (N=XX) | | | | | | | (N=XX) | ) | | | |
| | Mild | | Moderate | | Severe | | Mild | | Moderate | | Severe | : |
| | n (%) | nAE | n (%) | nAE | n (%) | nAE | n (%) | nAE | n (%) | nAE | n (%) | nAE |
| NUMBER OF SUBJECTS WITH AT | xx (xx.x) | XX | XX | XX | xx (xx.x) | XX | xx (xx.x) | XX | XX | XX | xx (xx.x) | XX |
| LEAST ONE AE | | | (xx.x) | | | | | | (xx.x) | | | |
| SOC1 | xx (xx.x) | XX | XX | XX | xx (xx.x) | XX | xx (xx.x) | XX | XX | XX | xx (xx.x) | XX |
| | | | (xx.x) | | | | | | (xx.x) | | | |
| PT1 | xx (xx.x) | XX | XX | XX | xx (xx.x) | XX | xx (xx.x) | XX | XX | XX | xx (xx.x) | XX |
| | | | (xx.x) | | | | | | (xx.x) | | | |
| PT2 | xx (xx.x) | XX | XX | XX | xx (xx.x) | XX | xx (xx.x) | XX | XX | XX | xx (xx.x) | XX |
| | | | (xx.x) | | | | | | (xx.x) | | | |
| PT3 | xx (xx.x) | XX | XX | XX | xx (xx.x) | XX | xx (xx.x) | XX | XX | XX | xx (xx.x) | XX |
| | | | (xx.x) | | | | | | (xx.x) | | | |
| SOC2 | xx (xx.x) | xx | XX | xx | xx (xx.x) | xx | xx (xx.x) | XX | XX | xx | xx (xx.x) | xx |
| | | | (xx.x) | | | | | | (xx.x) | | | |
| PT1 | xx (xx.x) | XX | XX | XX | xx (xx.x) | XX | xx (xx.x) | XX | XX | XX | xx (xx.x) | XX |
| | | | (xx.x) | | | | | | (xx.x) | | | |
| PT2 | xx (xx.x) | XX | XX | XX | xx (xx.x) | XX | xx (xx.x) | XX | XX | XX | xx (xx.x) | XX |
| | | | (xx.x) | | | | | | (xx.x) | | | |
| PT3 | xx (xx.x) | XX | XX | XX | xx (xx.x) | XX | xx (xx.x) | XX | XX | XX | xx (xx.x) | XX |
| | | | (xx.x) | | | | | | (xx.x) | | | |

N (%) = Number (percent) of subjects

nAE = Number of adverse events

Program file name xxxxxxxxxxxxxxxxxx

Programmer's note: Same format for table 9.4.4

Figure 9.3.3.1

Dermatologist Assessment Scores - Total Score
Safety Population



- \* = Significant difference from baseline (p < 0.05)
- # = Significant difference from baseline between groups

Programmers Note: Figure to be created for Safety population. Same format for figures 9.3.2.1 Change the title, footnote and time points to match protocol.

Listing 2.1 Adverse Events Safety Population

Product Group: Physiogel Calming Relief SPF 20 Cream

| Subject<br>Number | Age/<br>Sex/<br>Race[1] | Adverse Event<br>(Preferred<br>Term)<br>[System Organ | Start Date<br>(Study<br>Day)[2] | Start<br>Time | End Date | End<br>Time | Frequency/<br>Intensity[3] | Related<br>to Study<br>Product? | Action<br>Taken re<br>Study<br>Product | Outcome | Seri<br>ous? | With-<br>drew?<br>[4] |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|---|---|---|---|

PPD

Programmer's note: Same format for Listing 2.3.

<sup>@</sup> Subject excluded from the Safety Population.

<sup>[1]</sup> Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, O = Multiple.

<sup>[2]</sup> Study day is the day relative to start of treatment, day 1 being the day of first treatment.

<sup>[3]</sup> INT = Intermittent and SGLE = Single.

<sup>[4]</sup> Did subject withdraw from study as a result of this adverse event?

# Listing 2.2 Adverse Events Non-randomized Subjects

| Subject Age/ Adverse Event Start Date Start End Date End Frequency/ Related Number Sex/ (Preferred Time Time Intensity[2] to Study Race[1] Term) Product? [System Organ Class] | Action<br>Taken re<br>Study<br>Product | Outcome | Seri<br>ous? | With-<br>drew?<br>[3] |
|---|---|---|---|---|
|---|---|---|---|---|

PPD

<sup>[1]</sup> Age in years; Sex: F = Female, M = Male; Race: A = Asian, B = Black or African American, I = American Indian or Alaska Native, H = Native Hawaiian or Other Pacific Islander, W = White, O = Multiple.

<sup>[2]</sup> INT = Intermittent and SGLE = Single.

<sup>[3]</sup> Did subject withdraw from study as a result of this adverse event?

Listing 2.4
Randomization Details
All Randomized Subjects

| Subject Number | Age/Sex/Race [1] | Randomization Number | Randomized Treatment | Randomization Date |
|---|---|---|---|---|
| PPD | | | | |

[1] Age in years; Sex: F = Female, M = Male ; Race: A = Asian, B = Black or African American, I = American Indian or Alaska